CLINICAL TRIAL: NCT04560426
Title: Protective Effect of Intraoperative Parathyroid Gland Auxiliary Recognition System in Thyroid Malignant Tumor Operation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PTIOP1.0
Record Dates: First submitted 2020-08-29; First posted 2020-09-23 (Actual); Last update posted 2020-09-23 (Actual); Status verified 2020-09

CONDITIONS: Parathyroid; Intraoperative Monitoring; Thyroid Cancer
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Naked eyes & Instrument assistance (Experimental): Identify the parathyroid glands through the experience of surgeons and assistance of instrument.
  Interventions: Device: Intraoperative parathyroid gland auxiliary recognition system
- Naked eyes only (No Intervention): Identify the parathyroid glands only through the experience of surgeons.

INTERVENTIONS:
Device: Intraoperative parathyroid gland auxiliary recognition system — The enrolled patients are grouped according to whether or not to use the intraoperative parathyroid auxiliary recognition system.
  Arms: Naked eyes & Instrument assistance

SUMMARY:
This intraoperative parathyroid gland auxiliary recognition system uses the principle of parathyroid gland autofluorescence to assist surgeons in accurately identifying and protecting parathyroid glands during surgery, reducing the possibility of postoperative hypoparathyroidism. This study will explore the protective effect of the parathyroid gland auxiliary recognition instrument on parathyroid function during thyroid malignant tumor surgery through reasonable grouping.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with unilateral thyroid malignancies who require surgical treatment between the ages of 20-50.
2. No history of neck surgery and radiotherapy.
3. There is no evidence of parathyroid tumor invasion in preoperative imaging assessment.
4. No abnormal calcium metabolism disease.
5. No abnormalities in blood calcium and blood PTH before operation.
6. No allergy to contrast agents.
7. The patient or his agent signs an informed consent statement.

Exclusion Criteria:

1. Does not meet the entry criteria;
2. Parathyroid glands were found to be invaded by tumor during operation and the parathyroid glands could not be preserved.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-10-31 (Estimated); Primary Completion 2021-10-31 (Estimated); Study Completion 2022-10-31 (Estimated)

PRIMARY OUTCOMES:
Serum Calcium level | 24 hours after surgery
  Patients' serum Calcium level at 24 hours after surgery.
Serum Calcium level | 1 month after surgery
  Patients' serum Calcium level at 1 month after surgery.
PTH | 24 hours after surgery
  Patients' serum PTH level at 24 hours after surgery.
PTH | 1 month after surgery
  Patients' serum PTH level at 1 month after surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China